CLINICAL TRIAL: NCT03299751
Title: Evaluation of Biomarkers Combination Performance for the Diagnosis of Neonatal Sepsis in NICU Hospitalized Newborns
Brief Title: Evaluation of bioMarkErs to Reduce Antibiotics Use in hospitalizeD nEonates
Acronym: EMERAUDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 69HCL17_0492
Record Dates: First submitted 2017-09-28; First posted 2017-10-03 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Late-Onset Neonatal Sepsis
Keywords: neonatal sepsis; biomarker combination; diagnostic; antibiotic use; newborn; preterm neonates; NICU
MeSH Terms: conditions — Neonatal Sepsis; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- NICU newborns of at least 7 days of life with suggestive signs (Experimental)
  Interventions: Biological: Diagnostic performances of biomarkers combination

INTERVENTIONS:
Biological: Diagnostic performances of biomarkers combination — A blood sample of 400µL will be drawn at inclusion, when neonatal sepsis is suspected, at the same time of a venipuncture prescribed for standard care.
  The dosage of 11 biomarkers will be performed in a central laboratory. The adjudication committee composed with 3 neonatalogists will classify patients in 3 groups (infected, not infected or unclassified patients), based on their clinical and biological data obtained, through the standard of care practice, during the 48 hours following inclusion. The adjudication committee will be blinded to the biomarkers results.
  The adjudication committee composed with 3 neonatalogists will classify patients in 3 groups (infected, not infected or unclassified patientsconfirmed infection, refuted infection), based on their clinical and biological data obtained, through the standard of care practice, during the 48 hours following inclusion. The adjudication committee will be blinded to the biomarkers results.

SUMMARY:
Late-onset neonatal sepsis (LOS), occurring in newborn of at least 7 days of life, is frequently observed in Neonatal Intensive Care Units (NICUs) and potentially severe (mortality, neurologic and respiratory impairments).

Despite its high prevalence, a reliable diagnostic remains difficult. Currently, nonspecific clinical signs that might be linked to other neonatal conditions, such as prematurity and birth defects are used to determine the diagnosis of LOS. Laboratory results of biological markers, such as C-Reactive Protein (CRP) and Procalcitonin (PCT) are often delayed in comparison with LOS onset. Blood culture results are too late and lack sensitivity.

Excessive antibiotic use is observed in a large proportion of NICU hospitalized newborns. This results in an increased antibiotic resistance, microbiota modification, neonatal complications (pulmonary, ophthalmologic and neurologic) and mortality.

The primary objective is to identify, on a cohort of 250 patients, the optimal biomarker combination with good diagnostic performance (i.e. with maximal Area Under the ROC Curve) to early exclude a LOS diagnostic in newborns of at least 7 days of life with suggestive signs.

This identification will be carried out, as a secondary objective, with a sub-group of pre-term neonates whose birth weight is less than 1500 grams. The diagnostic value of the clinical signs that are suggestive of LOS will also be determined (sensitivity, specificity, negative and positive predictive values).

Once identified, the biomarker combination is expected to reduce unjustified antibiotic use.

ELIGIBILITY:
Inclusion Criteria:

* patients hospitalized in NICU;
* patients with suggestive signs of LOS including at least one of the following:

  o Fever > 38°C; tachycardia > 160bpm160 bpm; capillary refill time > 3 seconds; grey and/or pale skin complexion; apnea/ bradycardia syndrome,; bloating; rectal bleeding; hypotonia; lethargy; seizures without other obvious cause; increased ventilatory support and/or increased FiO2; cutaneous rash; inflammation at the needle-puncture site of the central venous catheter;
* patients with a standard of care blood sampling, including at least a blood culture;
* consent form signed by at least one parent/ legal representative.

Exclusion Criteria:

* patients treated with antibiotics for a bacteriologically confirmed infection at the moment of/ or 48 hours before blood sampling
* patients who underwent surgery during the 7 days prior to inclusion
* patients vaccinated during the 7 days prior to inclusion

Min Age: 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2020-11-20 (Actual); Study Completion 2020-11-20 (Actual)

PRIMARY OUTCOMES:
LOS diagnosis in NICU newborns of at least 7 days of life with suggestive clinical signs, confirmed by adjudication committee | hour 48
  The primary outcome measure will be determined by an independent adjudication committee that will classify the patients into the following categories: infected, not infected or unclassified patients. This committee will be blinded to the biomarkers that will be used to identify a combination with the best negative predictive value. It will be composed of two neonatologists and a pediatrician specialized in the child infectious diseases.
  The diagnostic performance of the biomarkers combination will be based on the adjudication committee

SECONDARY OUTCOMES:
LOS diagnosis in NICU preterm neonates, whose weight at birth is less than 1500 grams, of at least 7 days of life, with suggestive clinical signs, confirmed by adjudication committee. | Hour 48
  The primary outcome measure will be determined by an independent adjudication committee that will classify the patients into the following categories: infected, not infected or unclassified patients. This committee will be blinded to the biomarkers that will be used to identify a combination with the best negative predictive value. It will be composed of two neonatologists and a pediatrician specialized in the child infectious diseases.
  The diagnostic performance of the biomarkers combination will be based on the adjudication committee classification (gold standard).

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospices Civils de Lyon, Bron
  - CHU de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pons S, Trouillet-Assant S, Subtil F, Abbas-Chorfa F, Cornaton E, Berthiot A, Galletti S, Plat A, Rapin S, Trapes L, Generenaz L, Brengel-Pesce K, Callies A, Plaisant F, Claris O, Portefaix A, Flamant C, Butin M. Performance of 11 Host Biomarkers Alone or in Combination in the Diagnosis of Late-Onset Sepsis in Hospitalized Neonates: The Prospective EMERAUDE Study. Biomedicines. 2023 Jun 13;11(6):1703. doi: 10.3390/biomedicines11061703. PMID 37371798